CLINICAL TRIAL: NCT02578589
Title: Medial Plica Syndrome of the Knee: Conservative Treatment Versus Arthroscopic Plica Resection - a Randomized Controlled Multicenter Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regionshospitalet Silkeborg (Other)
Responsible Party: Principal Investigator, Steffen Sauer, Steffen Sauer, MD, Regionshospitalet Silkeborg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 280981PM
Record Dates: First submitted 2015-10-11; First posted 2015-10-19 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Plica Mediopatellaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery (Active Comparator)
  Interventions: Procedure: Plica resection vs conservative treatment
- Conservative treatment (Active Comparator)
  Interventions: Procedure: Plica resection vs conservative treatment

INTERVENTIONS:
Procedure: Plica resection vs conservative treatment — Plica resection vs conservative treatment

SUMMARY:
The purpose of this trial is to evaluate the effect of conservative treatment in comparison to arthroscopic resection of pathological medial plicae of the knee for patients with medial plica syndrome. The investigators expect conservative treatment to be significantly superior to arthroscopic plica resection with regard to symptom remission and return to prior functional level.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* History of antermedial knee pain
* Palpable medial band in clinical examination or medial plica appearence on MRI
* Absence of all of the following diagnoses: Osteoarthritis, osteochondritis dissecans, meniscal injury, patella subluxation, pes anserinus bursit, patellofemoral pain syndrome
* Given declaration of consent
* Joining a fitness centre for the duration of minimum 3 months at their own expense.

Exclusion Criteria:

Aged under 18 years

* Presence of one or more of the following diagnoses: Osteoarthritis, osteochondritis dissecans, meniscal injury, patella subluxation, pes anserinus bursit, patellofemoral pain syndrome
* Prior surgical intervention, infection, fracture or patellar luxation concerning the relevant knee
* Not willing to join a fitness centre for the duration of minimum 3 months at their own expense

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Lysholm-Scale (Units on a scale) | 2 years
  Difference of minimum 5 points concerning the average scoring outcome on the Lysholm Knee Scoring Scala in favor of patients undergoing conservative treatment in comparison to patients undergoing arthroscopic plica resection at 2 year follow up. Units of measure (Units on a scale)

SECONDARY OUTCOMES:
Kujala-Scale (Units on a scale) | 2 years
  Secondary endpoints: Higher average scoring outcome on the Anterior Knee Pain Scala (Kujala) in favor of patients undergoing conservative treatment in comparison to patients undergoing arthroscopic plica resection at 2 year follow up. Lower average results on Visual Anologue Scale concerning knee pain while walking indicated by patients undergoing conservative treatment in comparison to patients undergoing arthroscopic plica resection at 2 year follow up. Units of measure (Units on a scale)
QOL-Scale (Units on a scale) | 2 years
  Higher average scoring outcome on the Quality of Life Scala (extracted from KOOS) in favor of patients undergoing conservative treatment in comparison to patients undergoing arthroscopic plica resection at 2 year follow up. Units of measure (Units on a scale)
VAS-Scale (Visual Analog Scale for pain) (Units on a scale) | 2 years
  Lower average results on Visual Anologue Scale concerning knee pain while walking indicated by patients undergoing conservative treatment in comparison to patients undergoing arthroscopic plica resection at 2 year follow up. Units of measure (Units on a scale)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Regionshospital Silkeborg, Silkeborg
  - Regionshospitalet Silkeborg, Silkeborg